CLINICAL TRIAL: NCT00857181
Title: A Single-center, Open Study to Investigate Cytokine Levels in Patients With Hepatic Cirrhosis Before the Development of Significant Infection
Brief Title: Cytokines and the Risk of Infection in Liver Cirrhosis
Acronym: CLC-2009
Status: Terminated | Type: Observational
Why Stopped: Finding to be unable to reach the primary endpoint
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Vanessa Stadlbauer-Koellner, MD, MD, Medical University of Graz
Other Study IDs: CLC-2009-01
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; Infection; Inflammation; Cytokines
MeSH Terms: conditions — Liver Cirrhosis; Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver Cirrhosis: Single cohort of patients with liver cirrhosis to be investigated in the study. Two-monthly measurements of serum cytokines.

SUMMARY:
The aim of this study is to test whether the oscillation of cytokine concentrations in serum is able to predict the development of infection in patients with liver cirrhosis.

DETAILED DESCRIPTION:
Patients with liver cirrhosis frequently develop bacterial, viral or fungal infections which are the main trigger for decompensation of cirrhosis and development of complications and thereby infection hugely impacts morbidity and mortality in these patients. However, there is no clinical test available that allows rapid, on-site decision making if a patient is likely to develop an infection. The purpose of this study is to measure cytokines interleukin (IL) 6, IL8, IL10 and TNFalpha in patients with liver cirrhosis over a long follow-up period and test whether these inflammatory markers are able to predict the occurrence of infection before it becomes clinically significant. For this purpose, one hundred fifty consecutive patients with diagnosis of liver cirrhosis will be followed bi-monthly for 18 months. Blood samples will be collected for the cytokine measurements and infection cases will be reported at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical, radiological and/or histological evidence of liver cirrhosis
* Age above 18 (inclusive) at the time of screening
* Able and willing to give written informed consent and to comply with the requirements of the study

Exclusion Criteria:

* Infection during the last 14 days before screening
* Gastrointestinal bleeding within the last 14 days before screening
* Antibiotic therapy at the time of screening (except prophylaxis of spontaneous bacterial peritonitis)
* Shock or cardiac failure requiring inotrope treatment at the time of screening
* Hepatic encephalopathy grade >2
* Findings suggestive of organic nephropathy or a serum creatinine level of more than 2 mg/dl
* Human immunodeficiency virus infection at time of inclusion
* Use of immunomodulating agents within one month prior to screening (e.g. steroids)
* Any disease (e.g., advanced neoplasia) that could affect the short-term prognosis
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with biopsy proven or clinically evident liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Clinically significant infection requiring antibiotic, antiviral or antifungal treatment and hospitalisation. | 18 months

SECONDARY OUTCOMES:
All infections | 18 months
Hospitalisation for reasons other than infection | 18 months
Duration of hospitalisation | 18 months
Mortality | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD., Study Director — Medical University of Graz; Vanessa Stadlbauer-Koellner, MD., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria